CLINICAL TRIAL: NCT02209623
Title: Clinical Study of Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine (Tdap) Safety in Pregnant Women
Brief Title: TDAP Safety in Pregnant Women
Acronym: Tdap
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Duke University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathryn Edwards, Professor, Sarah Sell and Cornelius Vanderbilt Chair of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: CISA 2014 Task III
Record Dates: First submitted 2014-07-28; First posted 2014-08-06 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women receiving TDAP
  Interventions: Biological: TDAP

INTERVENTIONS:
Biological: TDAP

SUMMARY:
The purpose of this observational study is to evaluate the safety of Tetanus Toxoid Reduced Diphtheria, Toxoid, and Acelluar Pertussis Vaccine (Tdap) in pregnant women at ≥ 20 weeks 0 days gestation receiving Tdap as part of standard practice. Prior Tdap/Td/TT history will be verified by medical record review when possible. There will be an emphasis on enrolling women who have received Tdap before the current pregnancy, to the greatest extent possible. Non-pregnant women who are receiving their initial Tdap will also be recruited.

Injection-site (local) and systemic reaction data will be assessed on the vaccination day and during the 7 days following vaccination using either identical web-based or paper diaries, depending on the preference of the study participant.

Pregnant women will be followed until delivery with comprehensive obstetric and neonatal outcomes obtained from review of the electronic medical record.

DETAILED DESCRIPTION:
This is an observational study of both pregnant and non-pregnant women. Vaccine administration in the pregnant population will be part of routine care. Vaccine administration in the non-pregnant women will be provided as either routine care or as part of the study. Pregnant women at ≥ 20 weeks 0 days gestation who have not received Tdap during the current pregnancy will be enrolled, with prioritized emphasis on enrolling pregnant women who have received Tdap prior to the current pregnancy in order to attempt to address the question of closely-spaced repeated dosing. Detailed data will be collected from study participants on prior Tdap/Td/TT receipt. The non-pregnant women will consist of both Tdap naïve and those who have received Tdap previously. With Day 0 serving as the day of vaccination, participants will be followed through Day 7 for symptoms of reactogenicity. For Primary Objective 1, symptoms of reactogenicity occurring from Day 0 -7 will be compared between pregnant and non-pregnant women. For Objective 2, pregnant women will be followed through delivery for collection of pregnancy outcome data. Pregnancy outcomes among study participants will be compared with historical outcomes from summary data from both Vanderbilt and Duke. In addition, follow-up will be conducted for infants born to mothers who received Tdap during pregnancy to assess health outcomes and growth parameters through 6 months of life.

ELIGIBILITY:
Inclusion:

Subjects who meet the following criteria will be eligible to participate in this observational study. Tdap administration will be given as routine standard of care.

* Pregnant and non-pregnant women, as determined by medical history, aged 18 - 45 years of age inclusive
* For pregnant women only - Singleton gestation ≥ 20 weeks 0 days gestation - ≤34 weeks 0 days gestation based on reconciliation of last menstrual period and ultrasound dating. Estimated due date (EDD) and Gestational Age (GA) - EDD will be based on reconciliation of a "sure" first day of the last menstrual period (LMP) and earliest dating ultrasound. If the LMP is uncertain, then the earliest dating ultrasound will be used to determine EDD and GA. If the ultrasound derived-EDD is in agreement with sure-LMP derived EDD, then the LMP-derived EDD is used to determine GA. If the ultrasound derived EDD is not in agreement with the LMP-derived EDD, the ultrasound-derived EDD is used to determine GA.
* Intention of receiving Tdap vaccine based on ACIP guidelines
* Willing to provide written informed consent prior to initiation of any study procedures
* English or Spanish literate
* Intention of being available for entire study period and complete all relevant study procedures

Exclusion:

* Subjects who meet the following criteria will not be eligible to participate in this study:
* Febrile illness within the last 24 hours or an oral temperature > 100.4oF (> 38oC) prior to Tdap administration
* Severe allergic reaction (e.g., anaphylaxis) to any component of Tdap or any other diphtheria toxoid, tetanus toxoid and pertussis antigen containing vaccine
* Encephalopathy (e.g., coma, decreased level of consciousness, prolonged seizures) within 7 days of administration of a previous pertussis antigen-containing vaccine.
* Known or suspected impairment of immunologic function including active infection with HIV, hepatitis B or C, current use of glucocorticoids, i.e., oral, parenteral, and high-dose inhaled steroids, and immunosuppressive or cytotoxic drugs.
* Note, if a woman were to require antenatal corticosteroids for benefit of fetal lung maturity within 8 days post enrollment, she would not be excluded from the study for reactogenicity analysis. However, if antenatal corticosteroids were received anytime between vaccination and 28-day sample collection for serologic studies, she would be excluded from serologic studies as they could be altered by steroid receipt.
* Receipt of any licensed vaccine OR investigational product within 1 week prior to Tdap vaccination in this study or planning receipt of any vaccines during 8-day post-vaccination period.
* Note, any woman receiving an investigational vaccine or live vaccine inadvertently at any time during pregnancy will be excluded from analysis. (Note, inadvertent receipt of licensed HPV vaccine or any other inactivated licensed vaccine outside of the parameters specified above is not a reason for exclusion).
* Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.
* Anyone who is a relative of any research study personnel
* Anyone who is an employee of any research study personnel
* For pregnant women only
* Tdap/Td/TT receipt during current pregnancy prior to study enrollment
* Signs or symptoms of active preterm labor, defined as regular uterine contractions with cervical change
* For non-pregnant women only
* Intention of becoming pregnant during study participation
* Anyone who is already enrolled or plans to enroll in another clinical trial with an investigational product within 30 days of Tdap receipt. Co-enrollment in observational or behavioral intervention studies are allowed at any time while enrollment in a clinical trial involving an investigational product (other than vaccine) may occur after 30 days following Tdap receipt. Receipt of inactivated vaccines during pregnancy, including routinely recommended inactivated influenza vaccine, given as part of usual care, is not an exclusion for this study, except during the 8 days after Tdap vaccination

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 375 healthy pregnant women at ≥ 20 weeks 0 days gestation through ≤ 34 weeks 0 days gestation and their infants and 225 healthy non-pregnant women, age range 18-45 years
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Rates of injection-site and systemic reactions post Tdap administration. | 7 days post administration
  Rates of injection-site and systemic reactions after Tdap in pregnant women versus non-pregnant women will be compared.
Rates of preterm and small for gestational age (SGA) births in women who received Tdap prenatally | 7 days post delivery
  Rates of preterm and small for gestational age (SGA) births in women who received Tdap prenatally will be evaluated by review of the hospital delivery record following delivery.

SECONDARY OUTCOMES:
Differences in injection-site and systemic reactions in pregnant women who received Tdap before the current pregnancy versus women who are receiving their first Tdap dose | 7 days post vaccination
  Differences in injection-site and systemic reactions in pregnant women who received Tdap before the current pregnancy versus women who are receiving their first Tdap dose will be explored.
Rates of additional obstetrical and infant outcomes in pregnant women receiving Tdap | 7 days post delivery
  To assess rates of additional obstetrical and infant outcomes in pregnant women receiving Tdap including, but not limited to, maternal or fetal death, placental abruption, postpartum hemorrhage, pregnancy related hypertension, gestational diabetes
Health outcomes and growth parameters among infants born to women who received Tdap during pregnancy | 6 months post delivery
  To describe health outcomes and growth parameters through 6 months of life among infants born to women who received Tdap during pregnancy

OTHER OUTCOMES:
Measurement of serum cytokines before and after severe, local and systemic reactions | 28 days post vaccination
  Levels of cytokines will also be compared across groups (pregnant vs. non-pregnant women)
Measurement of serum antibody levels to pertussis toxin, filamentous hemagglutinin, pertactin, fimbria and diphtheria and tetanus toxins | 28 days post vaccination
  Antibody responses pre and post-vaccination will be compared between pregnant and non-pregnant women to each pertussis vaccine antigen

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Edwards, MD, Principal Investigator — Vanderbilt Medical Center; Geeta K Swamy, MD, Principal Investigator — Duke Medical Center; Karen R Broder, MD, Principal Investigator — Centers for Disease Control and Prevention; Kimberly B Fortner, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Duke University Dept of ObGyn, Division of Maternal-Fetal Medicine, Durham, North Carolina
  - Vanderbilt Medical Center, Vaccine Research Program, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortner KB, Swamy GK, Broder KR, Jimenez-Truque N, Zhu Y, Moro PL, Liang J, Walter EB, Heine RP, Moody MA, Yoder S, Edwards KM. Reactogenicity and immunogenicity of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Tdap) in pregnant and nonpregnant women. Vaccine. 2018 Oct 8;36(42):6354-6360. doi: 10.1016/j.vaccine.2018.07.012. Epub 2018 Sep 13. PMID 30219367